CLINICAL TRIAL: NCT04847791
Title: Lactoferrin for Treatment of Acute COVID-19 Infection in Hospitalized Patients: a Double-blind Multicenter Placebo-controlled Randomized Trial
Brief Title: Lactoferrin in Covid-19 Hospitalized Patients
Acronym: LAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paolo Manzoni (Other)
Responsible Party: Principal Investigator, Paolo Manzoni Study Group, MD, Paolo Manzoni
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020/279
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — coat protein, papaya mosiac virus

STUDY DESIGN:
Intervention Model Description: Prospective randomized double-blind placebo- controlled designed trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients are blind as Placebo administration consists of capsule identical with the same amount as an inert compound, starch of corn powder, and dispensed according to the same pattern of use. Care provider and investigator are blind as they do not know the capsule content (blisters are labelled: group 'A' or group 'B')
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Standard Anti-Covid-19 Therapy + Oral Administration of Bovine Lactoferrin 400mg (two capsules of Mosiac 200 product) every 12 h (i.e., fixed dose 800 mg / day) for 30 days and still away from meals
  Interventions: Dietary Supplement: Bovine lactoferrin
- Group B (Placebo Comparator): Standard anti-Covid-19 therapy + Placebo administration (capsule identical with the same amount as an inert compound, starch of corn powder), according to the same pattern of use.
  Interventions: Dietary Supplement: Placebo administration

INTERVENTIONS:
Dietary Supplement: Bovine lactoferrin — Oral Administration of Bovine Lactoferrin -fixed dose 800 mg / day for 30 days
  Other Names: MOSIAC
  Arms: Group A
Dietary Supplement: Placebo administration — capsule identical with the same amount as an inert compound, starch of corn powder), according to the same pattern of use.
  Arms: Group B

SUMMARY:
TRIAL LAC is a randomized double-blind non profit multicenter study with a nutritional product: bovine lactoferrin - Mosiac 200 mg.

the hypothesis to be confirmed is that bovine LF, administered daily orally in addition to standard therapies for 1 month to hospitalized patients with Covid-19 infection, can be useful to limit the severity, progression of the disease, shorten the time of swabs negativization (i.e. time required to eliminate the virus) and to reduce the morbidity load associated with it.

Patient recruitment will involve 2 centers in Italy: Ospedale degli Infermi (Ponderano, Biella) and AOU Maggiore della Carità (Novara).

The subjects enrolled will be randomized to two Groups:

Group A (experimental arm) - Standard Anti-Covid-19 Therapy + Oral Administration of Bovine Lactoferrin (fixed dose 800 mg / day) for 30 days Group B (control arm) - Standard anti-Covid-19 therapy + Placebo administration (identical capsule with the same amount as an inert compound, starch of corn powder), according to the same pattern of use.

It should be specified that the study treatment and placebo will be administered in addition to the standard care in place, and therefore in addition to all the pharmacological treatments currently used in clinical hospital practice against Covid-19.

DETAILED DESCRIPTION:
It has been shown with 'in vitro' studies that LF is able to prevent the entry of SARS-CoV-2 into the of the host cells.

Overall, the available evidence suggests that LF may be a therapeutic option that can be used to counteract and reduce the severity of Covid 19 infection. The study hase been designed in order to demonstrate efficacy of Lactoferrin in vivo.

Patients who will be admitted by Participating Centers for Covid-19 Infection will be screened for eligibility for study . If considered eligible, they will be offered participation in the Study, and it will be proposed and informed consent will be explained. Eligible patients will be registered in a centralized database at the IT systems of the University of Piedmont Orientale (UPO)/Hospital-University Company "Maggiore della Carità" of Novara. The pseudo-anonymized patient data will be recorded by the clinical centre in an 'ad hoc' Clinical Report Form with web-based access.

After obtaining informed consent, patients will then be randomised to LF or placebo group allocation using previous randomization lists Prepared. Randomization will take place on a competitive and balanced basis per clinical center participant. Permuted block randomization of size 4 will be implemented with an allocation ratio of 1:1 to ensure the balance between the groups of treatment. The randomization list will be managed through a REDCap randomization module.

The Hospital Pharmacy of the Participating Center, not involved in the enlistment of patients, will prepare a numbered sequence of sealed envelopes containing the code of allocation, and will keep its list that will remain inaccessible to the professionals involved in recruitment.These sealed envelopes will be opened sequentially, at the time of randomization.

The maintenance of the blind person will be guaranteed by keeping the staff randomization lists, i.e. the staff of the Hospital Pharmacy, on the one hand (staff who will also manage and deliver to the investigators the products being studied, which will look the same), and the randomizing and experimenting medical staff, on the other.

The logistical location of the two staff will also be completely separated, in sectors of the Hospital different and distant from each other, and not communicating in any way.

It should be pointed out that the patient enrolled by the clinical centers on the basis of the selection criteria can start standard-of-care therapy, in any case, before the randomization procedure being the identical basic therapeutic regimen in the two study arms.

For the calculation of the sample size required to demonstrate the primary endpoint, it was used a model built on historical data regarding the same endpoint. Pre-trial data from the two Participating Centres estimate the need for ICU admission at 25%; the need for mechanical ventilation in 30%; hospital mortality in 15%; the average duration hospitalization in 16 days.

The sample size was determined considering a two-sided t-test for two independent samples according to the following parameters:

1. A correct alpha level of 0.025 for two Bonferroni-method endpoints (Alpha total=0.025x2=0.05)
2. A total power of 0.8
3. A Cohen h effect size of 0.44 (corresponding to an effect standardized medium/small [Cohen 1977]), i.e. with a 14-day resignation rate of 60% for controls and 80% for treaties.

In this scenario, the size of the study achieved consists of 97 patients per arm of study. Calculations were performed using the R 3.6.1 software [Core Team 2015] and the pwr package [Champely 2018]. references:

* Cohen, J. Statistical power analysis for the behavioral sciences (rev.ed.1977).
* Core Team R: A Language and Environment for Statistical Computing; R Foundation for Statistical Computing: Vienna, Austria, 2015;
* Champely, S.; Ekstrom, C.; Dalgaard, P.; Gill, J.; Weibelzahl, S.; Anandkumar, A.;Ford, C.; Volcic, R.; De Rosario, H.; De Rosario, M.H. Package 'pwr.' R package version 2018, 1-2.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization in non-ICU ward for Covid-19 infection, with virological diagnosis SARS-CoV2 confirmed via RT-PCR (or quick test)
2. Age>18 aa
3. Covid symptomatology story from no more than 12 days

Exclusion Criteria:

1. Refusal of consent
2. Need for immediate admission to intensive care
3. Severe neoplasms (in advanced stage)
4. Allergies or intolerances known to Lactoferrin

4. Already being treated with Lactoferrin at the entrance to the Hospital 5. Patients with end-stage renal failure (stage 5) 6. Extremely serious general conditions to suggest an imminent exitus 7. Clinical conditions of absolute impossibility of tolerating ingestion of drugs/capsules due to conditions contraining the initiation of therapy for os.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
intensive care unit hospitalization rate | 1 year
  The primary endpoint will be to evaluate the efficacy of bovine LF orally (BLF- Mosiac) compared to placebo in affecting at least one of the following:
  1) it is expected a reduction of a composite event rate consisting of two items: the number of hospitalizations in intensive care unit due to any cause and the number of deaths
death | 1 year
  number of deaths during hospitalization
proportion of discharged patients | 1 year
  The primary endpoint will be to evaluate the efficacy of bovine LF orally (BLF- Mosiac) compared to placebo in affecting at least one of the following:
  2) it is expected an increase of proportion of discharged patients within 14 days and an increase of number of patients reaching a National Early Warning Score (NEWS) of 2 or less
National Early Warning Score (NEWS) | during hospitalization
  it is expected an increase of number of patients reaching a National Early Warning Score (NEWS) of 2 or less, maintained for at least 24hrs

SECONDARY OUTCOMES:
daily clinical severity score | during hospitalization
  Secondary Endpoints will be the assessment of a possible superiority of the experimental treatment compared to the standard treatment with regard to improving of the daily clinical severity score detected from the day of hospitalization to that of discharge and considering all the oucome hereafter listed
oxygen | during hospitalization
  the assessment of a possible superiority of the experimental treatment will be evaluated considering the need for additional oxygen (yes/no), and number of days of use
ferritin | during hospitalization
  lab values of ferritin
IL 6 | during hospitalization
  lab values of IL6
D dimers | during hospitalization
  lab vaules of D-dimers
hepcidine | during hospitalization
  lab vaules of hepcidine
ventilation | during hospitalization
  number of mechanical ventilation days (i.e., SIMV; SIPPV; HFOV etc) and/or CMO and number of days of ventilation in HFNC or CPAP
adverse events | during hospitalization
  registration of adverse events
pO2/FiO2 | during hospitalization
  it is expected achieving a value of pO2/FiO2 > 350 in two consecutive determinations, limited to the subgroup of patients in which this ratio was <300 at the entrance and in presence of radiologically and clinically documented pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Manzoni, MD, Principal Investigator — ASL BI
Locations (2):
- Italy (2):
  - ASL BI Ospedale degli Infermi, Ponderano, Biella
  - AOU Ospedale Maggiore della Carità, Novara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen JH, Jenssen H, Sandvik K, Gutteberg TJ. Anti-HSV activity of lactoferrin and lactoferricin is dependent on the presence of heparan sulphate at the cell surface. J Med Virol. 2004 Oct;74(2):262-71. doi: 10.1002/jmv.20171. PMID 15332275
- [Background] Avula A, Nalleballe K, Narula N, Sapozhnikov S, Dandu V, Toom S, Glaser A, Elsayegh D. COVID-19 presenting as stroke. Brain Behav Immun. 2020 Jul;87:115-119. doi: 10.1016/j.bbi.2020.04.077. Epub 2020 Apr 28. PMID 32360439
- [Background] Yang Z, Jiang R, Chen Q, Wang J, Duan Y, Pang X, Jiang S, Bi Y, Zhang H, Lonnerdal B, Lai J, Yin S. Concentration of Lactoferrin in Human Milk and Its Variation during Lactation in Different Chinese Populations. Nutrients. 2018 Sep 5;10(9):1235. doi: 10.3390/nu10091235. PMID 30189612
- [Background] Wang Y, Wang P, Wang H, Luo Y, Wan L, Jiang M, Chu Y. Lactoferrin for the treatment of COVID-19 (Review). Exp Ther Med. 2020 Dec;20(6):272. doi: 10.3892/etm.2020.9402. Epub 2020 Oct 27. PMID 33199997
- [Background] Wakabayashi H, Oda H, Yamauchi K, Abe F. Lactoferrin for prevention of common viral infections. J Infect Chemother. 2014 Nov;20(11):666-71. doi: 10.1016/j.jiac.2014.08.003. Epub 2014 Aug 30. PMID 25182867